CLINICAL TRIAL: NCT01539499
Title: Complications of Endocrine Surgery: Data From the United Health System Consortium
Brief Title: Complications of Endocrine Surgery: Data From the United HealthSystem Consortium
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 112685
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Thyroid Disease; Parathyroid Disease; Endocrine Gland
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to help better determine the complication rates for endocrine surgery across the nation for both benign and malignant disease. It is our hypothesis that the complication rates are low overall and that malignant disease results in a higher complication rate than benign disease. This study will do a database review from all University HealthSystem Consortium (UHC).

ELIGIBILITY:
Inclusion Criteria:

* All patients between the ages of 18 and 90 years who have a diagnosis of benign multinodular goiter and/or malignant thyroid disease and have undergone a total thyroidectomy as a primary procedure.
* Parathyroid patients will also be studied.

Exclusion Criteria:

* Non endocrine surgery patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted through a United HealthSystem Consortium query of endocrine surgery done as a primary procedure for specific diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Complication Rates for Endocrine Surgery | baseline
  The information presented in this report will provide a surgical tool for otolaryngologists to safely inform patients on the risks of endocrine surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Stack, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States